CLINICAL TRIAL: NCT02507921
Title: Comparing Type and Prevalence of HIV Drug Resistance in Treatment Experienced and naïve HIV-infected Adults in Uganda and Switzerland
Brief Title: Resistance in HIV+ in North and South
Acronym: RHINOS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Infectious Diseases Institute (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor-Investigator, Infectious Diseases Institute, Principal Investigator, Makerere University
Organization: Makerere University (Other)
Other Study IDs: ST/0112/15
Record Dates: First submitted 2015-06-16; First posted 2015-07-24 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: HIV Drug Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Plasma for HIV viral load and serum for storage
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators aim to assess type and frequency of HIV drug resistance in adults presenting to the Infectious Diseases Institute (IDI) in Kampala, Uganda, and compare this data to patients from the Swiss HIV Cohort Study (SHCS). This study is a single-site, cross-sectional study. The Investigators' goal is to perform viral load measurements in 2750 HIV-infected patients who have been on ART for 6 months or more. Presuming a detectable viral load in 10%, resistance testing would then be performed in 250 patients on ART. All adult patients attending will be screened for enrollment. Furthermore, the investigators' goal is to perform resistance testing in 250 ART naive patients in order to detect transmitted resistance mutations. Investigators will therefore consecutively screen and enroll 250 ART naive patients who attend the clinic during the study period. For each participant, a case report form (CRF) form will be completed which includes social, as well as medical information. Investigators will ask each participant for permission to store plasma in case resistance testing must be repeated, and serum, in case of future research questions.

DETAILED DESCRIPTION:
Background & Rational Uganda and Switzerland are two examples of regions in the world that have experienced the era of antiretroviral treatment (ART) in substantially different ways. While European patients had access to ART from the beginning of drug development, ART was made accessible to patients from sub-Saharan Africa many years later. HIV-infected patients in resource-limited settings were not subjected to the early days of treatment, were mono therapy was tried or combinations of drugs that are off the market nowadays. Furthermore, in contrast to European patients, patients from resource-limited settings were constantly confronted with economic constraints leading to stock-outs for instance. Cultural aspects, such as stigma and fear of disclosure, differ as well, and are well known to influence individual adherence and treatment outcome substantially.

Today similar first-line treatment choices are made by Ugandan and Swiss physicians, but monitoring strategies still differ. As in other countries of sub-Saharan Africa, treatment of HIV-infected patients is monitored immunologically and clinically, while viral load measurement is reserved for selected patients. In accordance with WHO recommendations treatment failure is therefore determined clinically (new or recurrent WHO stage III or IV condition) and/or by the decline of a patient's CD4 cell count to or below baseline, which usually occurs late during insufficient treatment. Viral rebound and emergence of resistance may thereby arise. Moreover, misclassification of treatment failure (e.g. patients with immunological failure in the absence of virological failure or complete non-adherence to treatment) may result in premature switching to more costly second-line treatment options.

The currently available information on transmitted drug resistance (TDR) in Ugandan adults shows lower rates compared to patients from European countries, including Switzerland. Yet, available studies were conducted with small patient numbers. Newer data from Uganda, especially under new WHO treatment recommendations, is not available yet.

To the best of investigators' knowledge, so far no study has directly compared HIV drug resistance data from a resource-limited country to a resource-rich country. Little is known about the effects of historically, culturally and economically different ART experiences on resistance. With the 2013 WHO guidelines, ART roll-out will be enhanced globally and the continued success of these large-scale treatment programs will depend on the prevention of further emergence of drug resistance.

Study Design:

Cross-sectional, single-site, observational Enrolment period: May 1st - July 31st 2015 Patients: All HIV-infected adults above the age of 18 years that have been on a stable first- or second-line ART regimen ≥6 months presenting to the Infectious Diseases Institute (IDI) during the study period and are able to give written informed consent will be enrolled. The goal is to perform viral load testing in 2750 patients on ART. Presuming a detectable viral load in 10%, resistance testing would then be performed in 250 patients on ART. Treatment naive HIV-infected patients above the age of 18 years presenting to the IDI during the study period will be offered resistance testing. The goal is to perform resistance testing in 250 ART naive patients.

Laboratory tests: A blood sample is used for resistance testing in treatment naive patients. For patients on ART, the initial sample will be used for HIV viral load measurement at the IDI. Part of the sample will be frozen (-80°C) and stored at the IDI for later resistance testing in case of detectable viral load (plasma viral load >1000 copies/ml). Resistance testing will be done at the Ugandan Virus Research Institute (UVRI) in Entebbe, Uganda.

Statistical Methods:

Type and frequency of mutations in treatment-naive will be identified and compared to the data from the SHCS. Investigators will compare treatment-naive patients from the SHCS who were tested in the same time-frame (in the year 2014). Additionally, investigators will identify a time-frame in the SHCS where a similar proportion of patients had detectable viral loads on ART as now in Uganda (the time-frame will depend on the findings in Uganda). Uni- and multivariate logistic regressions will be performed to identify risk factors for the detection of HIV drug resistance mutations.

Type and frequency of mutations in treatment-experienced patients will also be analyzed and compared to patients from the SHCS. For comparison, investigators will match patients from the SHCS with the same age, gender and ART. To identify risk factors for the detection of mutations in treatment-experienced patients, the investigators will also perform logistic regression models.

To study the diagnostic performance of clinical/immunological testing investigators will calculate the sensitivity, specificity, positive and negative predictive value compared to virological testing (gold standard).

These analyses will be performed for all drug-resistance mutations pooled together (outcome-variable= patient has any drug resistance mutation), for drug resistance mutations against individual drug classes (outcome = patient has any drug resistance mutation to a particular drug class), and for the two resistance mutations (M184V and K103N) that have been most prevalent in previous studies in resource-limited settings.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document indicating that the participant (or a legal representative) has been informed of all pertinent aspects of the study.
* Participants who are willing and able to comply with scheduled visits, laboratory tests, and other study procedures.
* Age ≥ 18 years
* ART naïve OR on stable ART regimen ≥ 6 months (first- or second-line)

Exclusion Criteria:

There are no exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be all HIV-1 infected adults presenting to the Infectious Disease Institute in Kampala during a defined study period, who are either treatment naïve or have been on a stable antiretroviral regimen for longer than 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 2750 (Estimated)
Dates: Start 2015-05; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
HIV drug resistance in treatment-naive patients | up to 12hrs
  Type and frequency of transmitted HIV drug resistance mutations detected in treatment naive patients and comparison to naive patients in the Swiss HIV Cohort Study (SHCS)
  • Identification of risk factors associated with the occurrence of transmitted HIV drug resistance mutations in treatment-naive patients
HIV drug resistance in treatment-experienced patients | up to 12hrs
  • Type and frequency of HIV drug resistance mutations detected in patients on ART with virological failure and comparison to patients on treatment the Swiss HIV Cohort Study (SHCS) Identification of risk factors associated with the detection of HIV drug resistance mutations in treatment-experienced patients

SECONDARY OUTCOMES:
Viroligical failure | up to 12hrs
  Proportion of HIV-infected patients with detectable viral load in the absence of immunological and/or clinical treatment failure
Viroligical failure | up to 12hrs
  • Diagnostic performance of immunological/clinical criteria for the detection of treatment failure compared to virological testing (gold standard)
Viroligical failure | up to 12hrs
  •Type and frequency of HIV drug resistance mutations detected in ART naive and experienced patients in Uganda and comparison to migrants from sub-Saharan Africa in the SHCS
Viroligical failure | up to 12hrs
  •Assessment of local risk factors for treatment failure

CONTACTS AND LOCATIONS:
Locations (1):
- Infectious Diseases Institute, Makerere University, Kampala, Uganda